CLINICAL TRIAL: NCT02355756
Title: Development of a Target Engagement Biomarker for Future PAC1 Antagonists With the Use of Intradermal Injected Maxadilan Induced Dermal Blood Flow Changes, Assessed by Laser Doppler Imaging
Brief Title: Biomarker Development for Future PAC1 Antagonists With Maxadilan
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCP14-3301-PAC1
Record Dates: First submitted 2015-01-15; First posted 2015-02-04 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — maxadilan protein, insect

ARMS (2):
- Active (Experimental): Intradermal injection of maxadilan solution
  Interventions: Drug: Maxadilan
- Placebo (Placebo Comparator): Intradermal injection of placebo (=vehicle) solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maxadilan
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
This will be a single center, open-label study in healthy male subjects between 18 and 45 years old to determine the dose response profiles of dermal blood flow in response to intradermal injections of maxadilan. The study will consist of 2 parts: Part I: dose and time finding and Part II: reproducibility over time.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a white male ≥18 and ≤ 45 years of age.
* Subject is a nonsmoker for at least 6 months prior to study start.
* Subject has a body mass index between 18-28 kg/m2.
* Subject is judged to be in good health on the basis of medical history, physical examination, vital signs, electrocardiogram, and routine laboratory data (including complete blood count, complete chemistry panel, prothrombin time and activated partial thromboplastin time (see Appendix C).
* Subjects must agree to practice a highly effective method of birth control during the study and for 1 week after dosing. Highly effective method of birth control includes sexual abstinence, vasectomy, or a condom in combination with hormonal birth control or intrauterine device (female partner).
* Subjects must agree not to donate sperm for the duration of the study.
* Subject understands the procedures and agrees to participate in the study by giving written informed consent.
* Subject agrees to refrain from strenuous physical activity 3 days before the screening visit, each study period and poststudy visit.

Exclusion Criteria:

* Subject has a history of any illness (including migraine) or has had/is expected to have surgery within 1 month of the start of the study which, in the investigator's opinion, might confound the results of the study.
* Subject has eczema, scleroderma, psoriasis, dermatitis, or keloids, tumors, ulcers, burns, flaps, or grafts on their forearm or other abnormality of the skin which may interfere with the study assessments.
* Subject has excessive hair growth on volar surface of the forearm.
* Subject cannot avoid excessive tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study and cannot cover forearms for 24 hours prior to each treatment period.
* Subject has a history of significant (drug) allergies including adverse experiences of a serious nature related to the administration of either a marketed or investigational drug or allergic reactions related to insect bites
* Subject currently uses any prescription or nonprescription drugs on a regular basis which cannot be discontinued for the duration of the study; subject has used any prescription or nonprescription medication within 14 days of the start of the study.
* Subject currently uses lotions, oils, depilatory preparations, or other topical treatments on the arms on a regular basis which cannot be discontinued for the duration of the study; subject has used any topical treatments within 7 days of the start of the study.
* Subject is a habitual and heavy consumer of coffee or caffeinated beverages (more than approximately 4 cups of tea, coffee, or cola drinks/day) at the time of the study. Subjects who have reduced their consumption to 4 cups of coffee/day at least 1 week prior to enrollment may participate. Subjects who cannot restrain from caffeinated beverages 12 hours before the study visit.
* Subject is unable to refrain from drinking alcohol 24 hours prior to maxadilan dosing, is currently a regular user (including "recreational use") of any illicit drugs, or has a history of drug (including alcohol) abuse.
* Subject has a positive urine drug test or alcohol breath test at screening or predose in period 1. The drug screens will include amphetamines / methamphetamines, methylenedioxymethamphetamine, benzodiaze-pines, barbiturates, cocaine, cannabis, tricyclic antidepressants, methadone and opiates.
* Subject is a smoker, cannot refrain from being around second hand smoke 24 hours prior to maxadilan dosing, or uses nicotine-containing products. Ex-smokers should have ceased smoking at least 6 months prior to screening. Nonsmokers will be confirmed by negative urinary cotinine tests at screening and predose period 1.
* Subject has any of the following vital sign measurements at screening: Heart Rate <40 or >100 beats/min, Diastolic Blood Pressure <50 or >89 mmHg, Systolic Blood Pressure <90 or >139 mmHg, Temperature <35 or >37.4 degrees Celsius, Respiration rate <7 or >25 R/min.
* Subject has any significant ECG abnormality.
* The subject has a positive prestudy human immunodeficiency virus-1/2 antibodies (HIV-1/2Ab), Positive Hepatitis B Surface Antigen (HepBsAg) (indicative of chronic Hepatitis B) or detectable Hepatitis C virus Ribonucleic acid (RNA) by Polymerase Chain Reaction (PCR) (indicative of active Hepatitis C - screening is generally done by Hepatitis C Antibody (HepCAb), followed by Hepatitis C virus RNA by PCR if HepCAb is positive) result at screening.
* Subject has been involved in testing an investigational drug in another clinical study within the last 4 weeks.
* Subject is in a situation or has a condition which, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in dermal blood flow induced by intradermal injections of maxadilan, compared to baseline and placebo for different doses, time point and in terms of reproducibility over time (i.e. inter-period reproducibility). | Every studyvisit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II)
Changes in vital signs. | Every studyvisit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II) and at 5-7 days after last studyvisit (post-study visit)
  as a measure of safety
Changes in ECG. | Every studyvisit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II) and at at 5-7 days after last studyvisit (post-study visit)
  as a measure of safety
Change in laboratory safety tests. | Every studyvisit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II) and at at 5-7 days after last studyvisit (post-study visit)
  as a measure of safety
Change in physical examination. | Every studyvisit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II) and at at 5-7 days after last studyvisit (post-study visit)
  as a measure of safety

SECONDARY OUTCOMES:
Tolerability of intradermal injections of maxadilan in healthy male subjects. Assessed using the Numerical rating scale-11 for pain. | Every study visit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II) and at at 5-7 days after last studyvisit (post-study visit)
  Assessed using the Numerical rating scale-11 for pain.
Change in dermal blood flow induced by intradermal injections of maxadilan, compared to baseline and placebo in terms of reproducibility between arms (i.e. inter-arm reproducibility. | Every studyvisit (Day 1, 8 and 15 for part I/Day 1 and 8 for part II)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Pharmacology, UZ Leuven, Leuven, Vlaams-Brabant, Belgium